CLINICAL TRIAL: NCT00098228
Title: Dose-Ranging Study in Patients With COPD
Brief Title: Dose-Ranging Study in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAB149B2205
Record Dates: First submitted 2004-12-03; First posted 2004-12-06 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: COPD
Keywords: COPD, adults, QAB149
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol

INTERVENTIONS:
Drug: QAB149

SUMMARY:
The trial is designed to identify an appropriate dose of QAB149 for delivery via a multiple dose inhaler for use in the COPD Phase III program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* Age 40-75 years
* Smoking history

Exclusion Criteria:

* Other serious disease
* Allergy to QAB149
* Respiratory tract infection

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 686 (Actual)
Dates: Start 2004-07; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Pulmonary function measured between 22 and 24 hours after dosing on Day 1

SECONDARY OUTCOMES:
Pulmonary function measured on days 1 and 7 at various intervals after dosing
Safety measurements

CONTACTS AND LOCATIONS:
Overall Officials: Novartis East Hanover — 862-778-8300
Locations (54):
- United States (54):
  - UAB Pulmonary Research, Birmingham, Alabama
  - Diagnostic & Medical Clinic, Mobile, Alabama
  - The University of South Alabama Medical Center, Mobile, Alabama
  - Pulmonary Associates, Phoenix, Arizona
  - USC Rancho Amigos Medical Center, Downey, California
  - Radiant Research, Encinitas, California
  - Allergy Research Foundation , Inc, Los Angeles, California
  - David Geffin UCLA School of Medicine, Los Angeles, California
  - Southern California Research, Mission Viejo, California
  - California Allergy & Asthma Medical Group, Palmdale, California
  - Allergy Associates Medical Group, Inc, San Diego, California
  - Allergy & Asthma Associates of Santa Clara Research Center, San Jose, California
  - Bensch Clinical Research Associates, Stockton, California
  - Rocky Mountain Center for Clinical Research, Wheat Ridge, Colorado
  - Physician's Research Center, Hartford, Connecticut
  - University of Miami School of Medicine, Miami, Florida
  - Crescent Clinical Research, Pensacola, Florida
  - Cordova Medical Center, Pensacola, Florida
  - USF Asthma, Allergy & Immunology, Clinical Research Unit, Tampa, Florida
  - University Medical Associates, LLP, Augusta, Georgia
  - Radiant Research - Atlanta West, Austell, Georgia
  - Sneeze, Wheeze & Itch Associates, LLC, Normal, Illinois
  - Asthma and Allergy Center of Chicago S.C., River Forest, Illinois
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Center for Clinical Research, Tauton, Massachusetts
  - ClinSite, Inc., Ann Arbor, Michigan
  - University of Michigan Health System, Ann Arbor, Michigan
  - Pulmonary Respiratory Institute of Southeast Michigan, Livonia, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - Minnesota Lung Center, Minneapolis, Minnesota
  - The Clinical Research Center, St Louis, Missouri
  - Creigton University, Omaha, Nebraska
  - Univ. of Nebraska Medical Center--Pulmonary Research, Omaha, Nebraska
  - New England Clinical Research, North Dartmouth, New Hampshire
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Pulmonary & Allergy Associates, Springfield, New Jersey
  - AAIR Reseach Center, Rochester, New York
  - University of Noth Carolina--Pulmonary Division, Chapel Hill, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Cloverdale Research Facility, Winston-Salem, North Carolina
  - Oklahoma Allergy and Asthma Clinic, Oklahoma City, Oklahoma
  - VA Medical Center, Oklahoma City, Oklahoma
  - Healthcare Research Consultants Inc., Tulsa, Oklahoma
  - River Road Medical Group, Eugene, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Low Country Lung and Critical Care, Charleston, South Carolina
  - Upstate Pharmaceutical Research, Simpsonville, South Carolina
  - Asthma & Allergy Res. Associates, Dallas, Texas
  - Central Texas Health Research, New Baunfels, Texas
  - Sylvana Research, San Antonio, Texas
  - Trinity Clinic Office of Research Admin., Tyler, Texas
  - Madrona Medical Group, Bellingham, Washington
  - Pulmonary Consultants, PLLC, Tacoma, Washington